CLINICAL TRIAL: NCT00189410
Title: Phase II Trial With Combination Chemotherapy Consisting of Pegylated Liposomal Doxorubicin (PLD) and Carboplatin in Malignant Gynecologic Tumour's
Brief Title: Combination Chemotherapy Consisting of Pegylated Liposomal Doxorubicin and Carboplatin in Malignant Gynecologic Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: MedServ. GmbH, Wiesbaden (Unknown); Essex Pharma GmbH (Industry)
Responsible Party: Gabriele Elser, MedServ. GmbH, Wiesbaden
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-GYN 3
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Cancer of the Ovary Treated as 2nd Line Therapy; Muellerian Mixed Tumours; Tumours of the Uterus; Cervical Cancers; Non-Epithelial Ovarian Tumours
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — liposomal doxorubicin; Carboplatin

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin and Carboplatin

SUMMARY:
Pegylated Liposomal Doxorubicin as well as Carboplatin have been showed efficacy in monotherapy as in combination therapy of gynaecologic tumours. As there is no common standard in the therapy of recurrent ovarian carcinoma, tumours of the uterus nor for non-epithelial ovarian tumours at time of designing of this study, this trial shall evaluate the new and well tolerated combination therapy consisting of Pegylated Liposomal Doxorubicin and Carboplatin.

DETAILED DESCRIPTION:
Aim of these study is the evaluation of combination chemotherapy in a patient subset with gynecologic tumours on regard to tolerance and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a gynecologic tumour [(non-epithelial ovarian tumour without germcell-tumours, tumours of the uterus (eg. Muellerian mixed tumours, Endometrial carcinomas, Uterus sarcoma, Cancer of the cervix)]
* Target or non-target lesion. Patients with epithelial ovarian carcinoma are qualified also if they have a CA 125 increase only.
* Patients with ovarian carcinoma must have completed a platin-containing chemotherapy more than 6 months at least. Patients with other malignancies could have prior chemotherapy, but must'nt
* Prior Radiotherapy less than 25% of haemapoietic system is allowed, but should have completed at least 6 weeks prior or registration
* Prior antitumoral hormone therapy, or specific immunotherapy is allowed, treatment have to be completed at least 3 weeks prior of registration
* All women with childbearing potential have to be a negative pregnancy test within 7 days of registration
* Perfomance Status 0-2 ECOG or more than 60% according to Karnofsky Index
* Estimated expectancy of life of more than 12 weeks
* adequate hematologic, renal and hepatic function according to following definitions: absolute Neutrophils >= 1,5 n/L Platelets >= 100 n/L Bilirubine <= 1,25 x ULN estimated glomerular filtration rate (Jelliffe) >= 60 ml/min
* Patients who have given their signed and written informed consent to participate in the trial
* Patients must be geographically accessible for treatment and follow

Exclusion Criteria:

* More than 2 prior chemotherapies (or Radio-Chemotherapies)
* active infection or concurrent severe medical problems unrelated to malignancy which would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy
* application of other cytotoxic or antitumoral agents during study period
* Patients with a history of seizure disorder or central nervous system disorders
* History of congestive heart failure (NYHA Classification > 2, even if medically controlled.
* History of clinical and electrocardiographically documented myocardial infarction within the last 6 months.
* History of atrial or ventricular arrhythmias (> LOWN II)
* Women who are pregnant or breast feeding
* Fertile women not using adequate contraceptive measures
* Patients who have used any investigational drugs within 30 days of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-06; Primary Completion 2005-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Tolerance
Response Rate mainly in malignant uterine tumours

SECONDARY OUTCOMES:
Time to Progression mainly in malignant uterine tumours
Overall Survival mainly in malignant uterine tumours

CONTACTS AND LOCATIONS:
Overall Officials: Andreas du Bois, MD PhD, Principal Investigator — AGO-OVAR, AGO Ovarian Cancer Study Group
Locations (19):
- Germany (19):
  - Medical Practice Dr. Klare, Berlin
  - Evangelisches Krankenhaus, Dept. of Gynecology & Obstetrics, Düsseldorf
  - Univerisity Hospital; Dept. of Gynecology & Obstetrics, Erlangen
  - University hospital, Dept. of gynecology & obstetrics, Essen
  - University hospital , Dept. gynecologic & obestretics, Frankfurt
  - University of Freiburg; Dept of Gynecology & Obstetrics, Freiburg im Breisgau
  - Ernst-Moritz-Arndt University, Dept. of Gynecology & Obstetrics, Greifswald
  - MH Hannover, Dept. of Gynecology & Obstetrics, Hanover
  - St. Vincentius Hospital, Dept. of Gynecology & Obstetrics, Karlsruhe
  - Univerisity Clinic Schleswig-Holstein, Campus Kiel, Dept. for gynecology & obstetrics, Kiel
  - Otto-von-Guericke Univerisity, Dept. of Gynecology & Obstetrics, Magdeburg
  - University hospital, Dept. of Gynecology & Obstetrics, Mainz
  - Phillips University, Clinic fo gynecology, gyn endocrinology and oncology, Marburg
  - University hospital Muenchen-Grosshadern, Dept. of gynecology & obstetrics, München
  - University Hospital TU Muenchen; Dept. of Gynecology & Obstetrics, München
  - Humaine Vogtlandklinikum; Dept. of gynecology & obstetrics, Plauen
  - University hospital, Dept. gynecology & obstetrics, Tübingen
  - Schwarzwald-Baar Klinikum Villingen, Dept. Gynecology, Villingen-Schwenningen
  - HSK, Dr. Horst Schmidt Klinik, Dept. of Gynecology & Gyn. Oncology, Wiesbaden

REFERENCES:
- [Background] Gropp M, du Bois A, Burges A, Meier W. Combination of Pegliposomal Doxorubicin (PLD) and Carboplatin in gynecologic tumors - An AGO Study Group Phase I/II trial. Int J Gycecol Cancer 2003:13 Suppl 1, p 112
- See also: Homepage of the AGO Ovarian Cancer Study Group — http://www.ago-ovar.de